CLINICAL TRIAL: NCT02834468
Title: A Multicenter Randomized Study of Dexamethasone Combined With Rituximab, Cyclosporin and Intravenous Immunoglobulin in the Management of Newly Diagnosed ITP Patients
Brief Title: DEX Combined With RTX, CSA and IVIG in the Management of Newly Diagnosed ITP Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Linyi People's Hospital (Other); Liaocheng People's Hospital (Other); Qingdao University (Other)
Responsible Party: Principal Investigator, Ming Hou, Prof., Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-2016-Combined Therapy
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Immune Thrombocytopenia
Keywords: Dexamethasone; Rituximab; Cyclosporin; Intravenous Immunoglobulin
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — resiniferatoxin; Immunoglobulins, Intravenous; Inosine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): DEX Combined With RTX, CSA and IVIG All patients are assigned to receive dexamethasone (given orally at a dose of 40 mg per day for 4 days), rituximab (given intravenously at a dose of 500mg once), cyclosporin (given orally at a dose of 2.5-3 mg/kg per day for 28 days) and intravenous immunoglobulin (given intravenously at a dose of 5g per month for 6 months) for the treatment of adults newly diagnosed ITP patients.
  Interventions: Drug: DEX Combined With RTX, CSA and IVIG

INTERVENTIONS:
Drug: DEX Combined With RTX, CSA and IVIG — The investigators are undertaking a multicenter trial of 100 primary ITP adult patients from 5 medical centers in China. All participants receive dexamethasone (given orally at a dose of 40 mg per day for 4 days), rituximab (given intravenously at a dose of 500mg once), cyclosporin (given orally at a dose of 2.5-3 mg/kg per day for 28 days) and intravenous immunoglobulin (given intravenously at a dose of 5g per month for 6 months) for the treatment of adults newly diagnosed ITP patients.
  Other Names: The combined therapy for ITP

SUMMARY:
The project was undertaken by Qilu Hospital, Shandong University in China. In order to report the efficacy and safety of dexamethasone combined with rituximab, cyclosporin and intravenous immunoglobulin in the management of newly diagnosed ITP patients.

DETAILED DESCRIPTION:
The investigators are undertaking a multicenter trial of 100 primary ITP adult patients from 5 medical centers in China. All participants receive dexamethasone (given orally at a dose of 40 mg per day for 4 days), rituximab (given intravenously at a dose of 500mg once), cyclosporin (given orally at a dose of 2.5-3 mg/kg per day for 28 days) and intravenous immunoglobulin (given intravenously at a dose of 5g per month for 6 months) for the treatment of adults newly diagnosed ITP patients.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Untreated hospitalized patients, may be male or female, between the ages of 18 -60 years.
3. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
4. Eastern Cooperative Oncology Group（ECOG）performance status ≤ 2.
5. Willing and able to sign written informed consent

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received high-dose steroids or [2] intravenous immunoglobulin transfusion(IVIG)in the 3 weeks prior to the start of the study.
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections. Severe medical condition (lung, hepatic or renal disorder) other than ITP. 4.Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)

5.Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.

6.Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.

7.Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response (Complete Response) | The time frame is up to 3 months per subject
  CR. A complete response (CR) was defined as a sustained (≥ 3 months) platelet count ≥ 100×10^9/L
Evaluation of platelet response (Response) | The time frame is up to 3 months per subject
  R. A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia.
Evaluation of platelet response (No Response) | The time frame is up to 3 months per subject
  NR.No response (NR) was defined as platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.
Evaluation of platelet response (relapses) | The time frame is up to 9 months per subject
  A relapses was defined as platelet count falls below 30×10^9/L or bleeding accrues after achieving R or CR.

SECONDARY OUTCOMES:
The number and frequency of therapy associated adverse events | up to 9 months per subject

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Medeot M, Zaja F, Vianelli N, Battista M, Baccarani M, Patriarca F, Soldano F, Isola M, De Luca S, Fanin R. Rituximab therapy in adult patients with relapsed or refractory immune thrombocytopenic purpura: long-term follow-up results. Eur J Haematol. 2008 Sep;81(3):165-9. doi: 10.1111/j.1600-0609.2008.01100.x. Epub 2008 May 27. PMID 18510702
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182